CLINICAL TRIAL: NCT00894582
Title: Prospective Measurements of Intra-Abdominal Volume and Pulmonary Function After Repair of Massive Ventral Hernias With the Components Separation Technique
Brief Title: Prospective Study of Ventral Hernia Repair
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Gregory A. Dumanian, M.D., Division of Plastic and Reconstructive Surgery, Northwestern University
Other Study IDs: 0678-010
Record Dates: First submitted 2009-05-05; First posted 2009-05-07 (Estimated); Last update posted 2009-05-07 (Estimated); Status verified 2009-05

CONDITIONS: Ventral Hernia
Keywords: massive ventral hernia; abdominal volume; pulmonary function; components separation; abdominal compartments syndrome
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Components separation hernia repair — Components separation is one method currently employed for repair of massive ventral hernias. In this study we simply measured the volume of patients' abdomen (who were already undergoing this surgery) as well as their pulmonary function both pre and postoperatively.

SUMMARY:
Immediate post-operative abdominal compartment syndrome is a feared complication after hernia repair in patients with a "loss of abdominal domain." Replacement of the viscera within an unyielding stiff abdominal wall may compromise the perfusion of the intestines, elevate the diaphragm, and interfere with ventilation. The components separation technique, used to repair these massive hernias, employs bilateral relaxing incisions in the external oblique muscle and fascia in order to approximate the rectus abdominis muscles in the midline. Reducing a large volume hernia into the abdominal cavity and primary closure of the abdominal wall should cause problems both with abdominal compartment pressure and with postoperative ventilation, but in the investigators' 13-year experience with over 250 cases, this has not been seen clinically, and the investigators sought to understand why. The investigators' hypothesis is that releasing the rectus muscles from the external obliques expands the intra-abdominal compartment, reclaims lost domain, and thus reduces abdominal pressure and respiratory problems. The investigators have previously reported increased abdominal volumes using the components separation technique in a retrospective series, but patients were not standardized for the collection of data, and no pulmonary function tests were obtained in that series (Hadad, in press). The purpose of this study was to prospectively analyze the effect of this surgical technique on abdominal volume and pulmonary function.

DETAILED DESCRIPTION:
With approval from the Institutional Review Board of Northwestern University, twenty-one patients with large ventral hernias were selected due to their large hernia size from a pool of 130 patients undergoing abdominal wall reconstruction from January 2007 to December 2008. No patients were excluded based on co-morbid conditions. One patient of the 21 selected was excluded because his preoperative CT scan that was performed at an outside institution was stored in an incompatible format for analysis. Another patient was excluded because it was decided intra-operatively that she could be repaired in a tension-free manner without components separation and was closed with mesh alone. Standard abdominal and pelvic CT scans and pulmonary function tests were performed immediately before hernia repair, and 3 months after repair. Pulmonary function tests were interpreted by blinded members of the Department of Pulmonology. Intra-operative peak airway pressure, bladder pressure, postoperative oxygen requirement, diagnosis of pneumonia, and any other cardio-respiratory complications were recorded on the remaining 19 patients. Routine patient demographics, clinical characteristics, postoperative course and incidence of recurrence were prospectively collected on all patients. Statistical analysis was performed in an intention-to-treat manner, using paired student's t-test where applicable.

ELIGIBILITY:
Inclusion Criteria:

* any patient with a large ventral hernia already scheduled to undergo ventral hernia repair with components separation technique

Exclusion Criteria:

* any patient unwilling to comply with pre-operative pulmonary function testing, or postoperative pulmonary function testing or postoperative one-time abdominal CT scan

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12

PRIMARY OUTCOMES:
Change in abdominal volume | 3 months following hernia repair

SECONDARY OUTCOMES:
Change in pulmonary function | 3 months following hernia repair

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Plastic and Reconstructive Surgery, Northwestern.edu, Chicago, Illinois, United States

REFERENCES:
- [Derived] Agnew SP, Small W Jr, Wang E, Smith LJ, Hadad I, Dumanian GA. Prospective measurements of intra-abdominal volume and pulmonary function after repair of massive ventral hernias with the components separation technique. Ann Surg. 2010 May;251(5):981-8. doi: 10.1097/SLA.0b013e3181d7707b. PMID 20395855